CLINICAL TRIAL: NCT05575765
Title: Clinical Validation of Multimodal Digestive Endoscopy in the Diagnosis of Colorectal Lesions
Brief Title: Clinical Validation of Multimodal Digestive Endoscopy
Status: Suspended | Type: Observational
Why Stopped: At present, this exploratory study has preliminarily achieved the set goals, and the subsequent data analysis is currently underway to determine whether it is necessary to continue recruiting participants.
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Kaichun Wu, vice president, Xijing Hospital of Digestive Diseases
Other Study IDs: XijingMDERC
Record Dates: First submitted 2022-09-30; First posted 2022-10-12 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Neoplasms; Confocal Laser Endomicroscopy; Endoscopy, Digestive System; Molecular Imaging
Keywords: Probe-based confocal laser endomicroscopy; Endoscopic cerenkov luminescence imaging; Multimodal digestive endoscopy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with a clinical diagnosis of colorectal cancer, colorectal polyps, and colorectal adenomas

SUMMARY:
According to the latest global cancer epidemiological data published by the International Agency for Research on Cancer, colorectal cancer (CRC) ranks 3rd in total incidence and 2nd in total mortality among all malignancies worldwide. The prognosis of CRC is directly related to tumor stage. The 5-year survival rate for early CRC can reach 90%, while less than 14% for advanced CRC. Therefore, early diagnosis of CRC is particularly important. Gastrointestinal (GI) endoscopy is an important method in the diagnosis of CRC. Currently, diagnosis of GI endoscopy is mainly based on morphological changes of tumors, while early-stage tumors are difficult to be detected because of the indistinguishable morphology. Studies have shown that the molecular function of cancer cells can be altered in early-stage tumors. The development of a new endoscopic system that can identify early tumor molecular function changes and improve the accuracy of morphological diagnosis will greatly improve the early diagnosis rate of CRC, which is the future direction of GI endoscopic system design and development.

The combination of high-definition white light endoscopy, endoscopic cerenkov luminescence imaging (ECLI) and probe-based confocal laser endomicroscopy (pCLE) is ideal for future new GI endoscopy. High-definition white light endoscopy is helpful to quickly find and locate suspected abnormal mucosa; on top of this, ECLI enables molecule-specific functional imaging for accurate identification and determination of GI lesions; and further relies on pCLE for high-precision "cellular-level" lesion images for optical biopsy of lesions. Through the multimodal digestive endoscopy, structural imaging and functional imaging can be accomplished simultaneously, playing the innate advantage of multimodal information fusion diagnosis and facilitating the identification of early-stage tumors.

In this clinical trial, patients with colorectal lesions who underwent PET-CT in Xijing Hospital were enrolled. Multimodal digestive endoscopy, combination of high-definition white light endoscopy, ECLI and pCLE, was used to perform for each patient's colorectal lesion. ECLI images were compared with PET-CT images, and pCLE images were compared with lesion histopathology, which evaluate the actual imaging effect of multimodal digestive endoscopy in human.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years old.
2. Clinical diagnosis of colorectal cancer, colorectal polyps, colorectal adenomas and enteritis.
3. No allergy to relevant imaging agents.
4. Person who is able to understand and sign the informed consent form.
5. Person who is willing to participate in this experiment.

Exclusion Criteria:

1. Patient who has been treated for colorectal lesions (endoscopic treatment, surgery , targeted therapy, and radiotherapy, etc.)
2. Patients with severe, progressive, or uncontrolled diseases of the kidneys, liver, blood, gastrointestinal tract, endocrine system, lungs, heart, or nervous system.
3. Women who are pregnant or breastfeeding.
4. Person without personal freedom and independent civil capacity.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: grade III A hospital
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-11-11 (Actual); Primary Completion 2025-04-10 (Estimated); Study Completion 2025-04-10 (Estimated)

PRIMARY OUTCOMES:
The concordance rate between the results of multimodal digestive endoscopy for the diagnosis of early colorectal malignancies and the histopathological results | White light endoscopy takes 1 second; endoscopic cerenkov luminescence imaging takes 5 minutes; probe-based confocal laser endomicroscopy takes 2 minutes

SECONDARY OUTCOMES:
The concordance rate between the results of endoscopic cerenkov luminescence imaging for the diagnosis of early colorectal malignancies and the histopathological results | Endoscopic cerenkov luminescence imaging time: 1-5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Wu kaichun, PhD, Study Director — Xijing Hospital of Digestive Diseases
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen X, Wang X, Yan T, Zheng Y, Cao H, Ren F, Cao X, Meng X, Lu X, Liang S, Wu K. Sensitivity improved Cerenkov luminescence endoscopy using optimal system parameters. Quant Imaging Med Surg. 2022 Jan;12(1):425-438. doi: 10.21037/qims-21-373. PMID 34993091
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Schillaci O, Scimeca M, Toschi N, Bonfiglio R, Urbano N, Bonanno E. Combining Diagnostic Imaging and Pathology for Improving Diagnosis and Prognosis of Cancer. Contrast Media Mol Imaging. 2019 Jul 1;2019:9429761. doi: 10.1155/2019/9429761. eCollection 2019. PMID 31354394
- [Background] Moghbeli M. MicroRNAs as the critical regulators of Cisplatin resistance in ovarian cancer cells. J Ovarian Res. 2021 Sep 30;14(1):127. doi: 10.1186/s13048-021-00882-1. PMID 34593006
- [Background] Fan X, Qin X, Zhang Y, Li Z, Zhou T, Zhang J, You W, Li W, Pan K. Screening for gastric cancer in China: Advances, challenges and visions. Chin J Cancer Res. 2021 Apr 30;33(2):168-180. doi: 10.21147/j.issn.1000-9604.2021.02.05. PMID 34158737
- [Background] Luu XQ, Lee K, Jun JK, Suh M, Jung KW, Choi KS. Effect of gastric cancer screening on long-term survival of gastric cancer patients: results of Korean national cancer screening program. J Gastroenterol. 2022 Jul;57(7):464-475. doi: 10.1007/s00535-022-01878-4. Epub 2022 May 14. PMID 35568752
- [Background] Hamashima C, Goto R. Potential capacity of endoscopic screening for gastric cancer in Japan. Cancer Sci. 2017 Jan;108(1):101-107. doi: 10.1111/cas.13100. Epub 2016 Dec 12. PMID 27727490
- [Background] Cao X, Chen X, Kang F, Lin Y, Liu M, Hu H, Nie Y, Wu K, Wang J, Liang J, Tian J. Performance evaluation of endoscopic Cerenkov luminescence imaging system: in vitro and pseudotumor studies. Biomed Opt Express. 2014 Sep 17;5(10):3660-70. doi: 10.1364/BOE.5.003660. eCollection 2014 Oct 1. PMID 25360380
- [Background] Hu H, Cao X, Kang F, Wang M, Lin Y, Liu M, Li S, Yao L, Liang J, Liang J, Nie Y, Chen X, Wang J, Wu K. Feasibility study of novel endoscopic Cerenkov luminescence imaging system in detecting and quantifying gastrointestinal disease: first human results. Eur Radiol. 2015 Jun;25(6):1814-22. doi: 10.1007/s00330-014-3574-2. Epub 2015 Jan 11. PMID 25577521
- [Derived] Yang Z, Wu Z, Pang T, Liu D, Wang X, Yu J, Xu S, Kang X, Liao D, Tian Z, Bai Y, Xi X, Yan T, Lu X, Qi Y, Zhang M, Zhao L, Kang F, Liang S, Wang J, Chen X, Wu K. Early diagnosis of colorectal cancer using Cerenkov luminescence endoscopy: a pilot trial involving humans for the first time. Theranostics. 2026 Jan 8;16(7):3685-3696. doi: 10.7150/thno.122007. eCollection 2026. PMID 41608582